CLINICAL TRIAL: NCT06907771
Title: Study of the Impact on Survival of a Paradigm Shift in the Therapeutic Strategy of Patients With Advanced Ovarian Cancer
Acronym: PACO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9301
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ovarian cancer is the 8th leading cause of cancer-related death in women. Its prognosis is poor, with diagnosis often made at an advanced stage.

Patient management has evolved in recent years with more radical surgeries and the introduction of maintenance treatment following neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Operated on at the HUS between January 1, 2010 and December 31, 2022
* Having undergone primary or interval cytoreductive surgery
* Suffering from stage FIGO IIIC or IV high-grade serous carcinoma of ovarian origin

Exclusion Criteria:

* Patiente ayant exprimé son opposition à la réutilisation de ses données à des fins de recherches scientifiques.
* Autres types histologiques de cancer de l'ovaire
* Stades de la maladie FIGO I, II, IIIA et IIIC
* Chirurgie de clôture.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) having undergone primary or interval cytoreductive surgery
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Study of progression-free survival at 36 months | At 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gynécologique et d'Obstétrique - CHU de Strasbourg - France, Strasbourg, France